CLINICAL TRIAL: NCT03208296
Title: A Phase 1b/2a Study of ASN-002 to Treat Basal Cell Carcinomas (BCCs) in Individuals With Basal Cell Nevus Syndrome (BCNS)
Brief Title: Study of ASN-002 to Treat Basal Cell Carcinomas (BCCs) in Individuals With Basal Cell Nevus Syndrome (BCNS)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study did not start. Another protocol is being developed. Recruitment on hold.
Sponsor: Ascend Biopharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASN-002-002
Record Dates: First submitted 2017-06-29; First posted 2017-07-05 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Basal Cell Carcinoma in Basal Cell Nevus Syndrome
Keywords: Basal Cell Nevus Syndrome; Basal Cell Carcinoma
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Carcinoma, Basal Cell | interventions — gusacitinib

STUDY DESIGN:
Intervention Model Description: This is a dose escalation study to determine the safety and efficacy of ASN-002 in treatment of BCCs in BCNS patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Subjects with 4 or more lesions will receive 1.0 x 10^11 vp/injection of ASN-002 into each of 4 BCCs, weekly x 3, i.e. weeks 1, 2, and 3
  Interventions: Biological: ASN-002
- Cohort B 1.5 (Experimental): Subjects with 4 or more lesions will receive 1.5 x 10^11 vp/injection of ASN-002 into each of 3 BCCs, weekly x 3, i.e. weeks 1, 2, and 3
  Interventions: Biological: ASN-002
- Cohort B 1.0 (Experimental): Subjects with 4 or more lesions will receive 1.0 x 10^11 vp/injection of ASN-002 into each of 3 BCCs, weekly x 3, i.e. weeks 1, 2, and 3
  Interventions: Biological: ASN-002

INTERVENTIONS:
Biological: ASN-002 — ASN-002 has been designed for clinical applications, especially for intratumoral administration in the treatment of various cancers. This rAd vector delivers the gene of interest, in the case of ASN-002 the human IFNγ gene, into target cells. The rAd vector in ASN-002 is replication deficient and although it infects cells, it is not able to replicate in the tumor or in normal human cells. The infected cells are able to transcribe and translate the IFNγ DNA leading to a sustained local concentration of IFNγ in the tumor mass that is designed to avoid high levels of systemic IFNγ that may be lead to unacceptable toxicity.

SUMMARY:
The primary objective is to confirm the safety of treating multiple BCCs once weekly x 3 weeks in individuals with Basal Cell Nevus Syndrome (BCNS).

The secondary objectives of the study are to obtain preliminary data on the effectiveness of ASN-002 in the treatment of BCCs in individuals with Basal Cell Nevus Syndrome (BCNS) by

1. evaluating the histological clearance of BCCs in patients with BCNS, and
2. assessing the clinical changes of BCCs after treatment with ASN-002, and
3. assessing the systemic effect of ASN-002 by determining response in non-injected lesions
4. assess the safety and clinical changes after a second cycle of ASN-002 injections

DETAILED DESCRIPTION:
Methodology:

Patients with BCNS who meet the Eligibility Requirements below will be studied. After informed consent is obtained and baseline evaluation, each lesion to be injected will receive ASN-002 once weekly x 3 weeks. Subjects will be premedicated with acetaminophen, 1000mg, 30 minutes prior to injection and continue 650mg, four times/day for two days after injection. Evaluation for toxicity and safety will be performed at 1, 2, 3 and 4 months after the first injection. All target lesions will be excised at 6 months and the subject evaluated for healing one month later.

Subjects with 5 or more lesions will be entered into Cohort A and will receive 1.0 x 1011 vp/injection into each of 4 BCCs, weekly x 3, i.e. weeks 1, 2, and 3, i.e. a total dose of 4.0 x 1011 vp on each day of injections. If one subject in this cohort experiences Grade 3 or greater local or systemic toxicities by week 4, three additional subjects will be accrued to this cohort. If none of the first 3 subjects or no more than one of the six subjects in the expanded cohort experiences Grade 3 or greater local or systemic toxicities by week 4, the total dose of 4.0 x 1011 vp/day will be accepted for further clinical assessment. All four injected lesions and 1 or 2 non-injected lesions will be excised after 6 months.

Cohort B will be open for accrual to patients with 4 or more lesions once Cohort A is accepted for further clinical assessment or if Cohort A has >1/6 Grade 3 AEs. Subjects in Cohort B will receive 1.5 or 1.0 x 1011 vp/injection into each of 3 BCCs, weekly x 3, i.e. weeks 1, 2, and 3, i.e. a total dose of 4.5 or 3.0 x 1011 vp on each day of injections as outlined in Synopsis Table 2 below. If one subject in this cohort experiences Grade 3 or greater local or systemic toxicities by week 4, three additional subjects will be accrued to this cohort. If none of the first 3 subjects or no more than one of the six subjects in the expanded Cohort B1.5 or B1.0 experiences Grade 3 or greater local or systemic toxicities by week 4, that total dose of 4.5 or 3.0 x 1011 vp/day will be accepted for further clinical assessment. All three injected lesions and 1-2 non-injected lesions will be excised after 6 months.

Cohort C may be designed based on the results observed in Cohorts A and B with the agreement of the Protocol Steering Committee. If a total dose >4.5 x 1011 vp/day of injection ASN-002 on any single day or more than 3 weekly injections are to be administered, a formal amendment to the Protocol must be approved before accrual to Cohort C is permitted.

Each cohort will be assessed for safety, dose escalation and possible cohort expansion as described above. The week 4 assessment of toxicity and apparent efficacy of the first 3 subjects in each cohort will be used to determine the need to increase the size of that cohort to 6 subjects. Cohorts will be assessed clinically at 1, 2, 3 and 4 months. Treated tumors will be resected at 6 months, based on observations in the ongoing Australia trial study that inflammation persisting at 16 weeks could not be reliably distinguished from residual tumor. The 1st and 3rd secondary endpoints, histological clearance of injected and non-injected lesions, will be assessed by the Pathology Department of each clinical site. Representative slides will be submitted for possible central review to be performed at the discretion of Ascend. Each participant will also be seen one month after tumor resection to assess healing and post-surgical results Each subject may be evaluated on the 7 month visit for a second cycle of 3 weekly ASN-002 injections into new or previously untreated BCC lesions at a dose accepted for further clinical assessment. Subjects who receive a second cycle will be followed for 6 months as before, but lesion excision will be at the discretion of the investigator.

In the event study subjects in any Cohort do not proceed to histological confirmation of response per protocol, they may be replaced as long as the reason for not proceeding to histological confirmation of response per protocol was not investigational product related adverse events and so long as the Protocol Steering Committee concurs with the Sponsor that no limiting safety issues have been identified.

Depending on results, and at the discretion of the Sponsor and the Protocol Steering Committee, one Cohort may be expanded to a total of 24 subjects so long as no more than one of six subjects already included at that dose and schedule of ASN-002 experienced Grade 3 or greater local or systemic toxicities. The selection of the cohort to be expanded will be based on favorable response data from the subjects already included at that dose and schedule of ASN-002,

ELIGIBILITY:
Inclusion Criteria:

1. Must satisfy established criteria for the diagnosis of BCNS (Section 1.1.2, Table 1).
2. Must have at least 4 target lesions, clinically consistent with BCC.
3. Up to 6 target lesions, including each of the 3 or 4 to-be-injected lesions and 1 or 2 non-injected lesions must be biopsied.
4. At least 3 target lesions, 2 to be injected and one to be non-injected, must be biopsy proven BCC per criteria in Synopsis Table 3: Modified Criteria for Low Risk BCC in BCNS Patients
5. Removal of < 25% of the area of the tumor by initial biopsy performed within 12 weeks before screening visit. A 2mm punch biopsy is recommended for histological confirmation of BCC.
6. Screening laboratory values as follows:

   1. Neutrophil count > 1500/mm3
   2. Hemoglobin > 10 g/dL
   3. Platelet count > 100,000/mm3
   4. Total bilirubin < 1.5 X upper limit of normal (ULN), except in the case of known Gilbert's syndrome
   5. Aspartate transaminase (AST), alanine transaminase (ALT) or alkaline phosphatase (ALP) < 1.5X ULN
   6. Creatinine < 1.5 X upper limit of normal (ULN)
7. 18 years of age or older at Screening visit.
8. Infertile, postmenopausal, surgically sterile or using acceptable and highly effective birth control methods for the duration of the study and for 3 months after last administration of ASN-002.
9. Written informed consent prior to initiation of study-specified procedures.
10. Able and willing to comply with all study requirements, including surgical removal of tumor/tumor sites as required by the study.

Exclusion Criteria:

1. Target tumor biopsy shows evidence of:

   * micronodular features,
   * squamous metaplasia,
   * sclerosing BCC,
   * morpheic BCC, or
   * peri-neural involvement.
   * cystic BCC
2. Eastern Cooperative Oncology Group (ECOG) performance status > 2.
3. Known or suspected metastatic disease.
4. Female participants must be non-lactating and non-pregnant.
5. Clinically active or uncontrolled skin disease that would interfere with evaluation of the area surrounding the target tumor (e.g. eczema, unstable psoriasis, xeroderma pigmentosa).
6. Known history of sensitivity to any of the ingredients in ASN-002.
7. Immunocompromised (e.g. known hepatitis B or C or HIV infection) or is receiving or is expected to receive an immunomodulating agent (including immunosuppressive agents, cytotoxic drugs, biological agents, immunoglobulins, interferon or other immune or cytokine-based therapies; regular use of inhaled or oral corticosteroids at doses higher than replacement doses is an exclusion criterion).
8. Treatment with psoralen plus UVA or UVB therapy within 3 months of screening and agrees not to receive such treatment until excision site is confirmed to be well healed at the post-surgery study visits
9. Prior systemic or local treatment for target tumors.
10. History of immunological disorder, severe allergic reaction, moderate or severe asthma or known history of anaphylaxis or any other serious adverse reactions to any medication.
11. Any serious or active medical or psychiatric illness or recreational or therapeutic drug or alcohol use that, in the opinion of the Investigator, would interfere with treatment, assessment or compliance with the protocol, or subject safety.
12. Any experimental or investigational agents within 1 month of first injection.
13. Any prior exposure to TG1041, TG1042 (ASN-002), any other adenoviral-based experimental agent within 5 months prior to screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety of ASN-002 will be studied in terms of AEs reported in individuals with Basal Cell Nevus Syndrome (BCNS) receiving ASN-002 using CTCAE 4.03. | The assessment will be conducted at every visit after first dose, week1, week2, week 3, Months1, 2, 3, 4 and at Month 6.
  Clinical safety will assessed in terms of changes in vital signs, AEs, serious AEs (SAEs), laboratory abnormalities and withdrawals from study. Local skin and injection site reactions will be assessed in detail scoring erythema, ulceration, pain and overall severity as none, mild, moderate or severe using protocol-specific modifications of the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

SECONDARY OUTCOMES:
Treatment efficacy in term of percentage of histological cure of BCC lesions at 6 months | 6 months from baseline
  At the end of the study, BCC lesions will be excised and studied under microscope to study the complete cure of BCC i.e. histological clearance
Clinical changes in BCCs after treatment with ASN-002 in- terms of change in lesion size (mm) | 6 months from baseline.
  The BCC lesions will be measured in mm at baseline, after first dose at Months1, 2, 3, 4 and at Month 6 to study the change in lesion size and clinical response.
The systemic effect of ASN-002 will be assessed for non-injected lesions by studying the change in lesion size from baseline to end of the study. | 6 months from baseline
  The non-injected BCC lesions will be measured in mm at baseline, after first dose at Months1, 2, 3, 4 and at Month 6 to study the change in lesion size and clinical response.
The safety in terms of the AEs reported (using CTCAE 4.03) after 6 months from first dose in retreatment cycle | 6 months
  Clinical safety will assessed in terms of changes in vital signs, AEs, serious AEs (SAEs), laboratory abnormalities and withdrawals from study. Local skin and injection site reactions will be assessed in detail scoring erythema, ulceration, pain and overall severity as none, mild, moderate or severe using protocol-specific modifications of the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
The systemic effect of ASN-002 will be assessed for non-injected lesions by studying the rate of histological clearance after 6 months of first dose. | 6 months from baseline
  At the end of the study, BCC lesions will be excised and studied under microscope to study the complete cure of BCC i.e. histological clearance
The efficacy will be assessed in terms of change in lesion size (mm) after 6 months from first dose in retreatment cycle | 6 months
  The change in lesions size in mm will be studied after 6 months from first dose in retreatment cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Leong, Study Chair — Ascend Biopharmaceuticals Ltd; Anna Bar, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be taken in due course of time.